CLINICAL TRIAL: NCT01735838
Title: Intrathoracic Bloodvolume Measurement by Contrast Enhanced Ultrasound: Validation of the Technique and Evaluation as a Measurement of Response to Cardiac Resynchronization Therapy: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Ingeborg Herold, MD, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL39385.060.12
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Intrathoracic Blood Volume in Heart Failure Patients

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Summary Rationale: Cardiac resynchronisation therapy (CRT) with biventricular pacemakers and implantable cardiac defibrillators (ICD) has proven to be a valuable therapy in selected patients with systolic heart failure, ameliorating both morbidity and mortality. However, with current selection criteria and implant technique, about 20 to 30 % of patients remain non-responders. Non-responders might be due to failing selection criteria or methodology in casu echocardiography. Moreover, the definition of response to CRT is unequivocal and there is a need for a simple and reproducible measure of response with low inter- and intra-observer variability.

Primary objectives: This study evaluates the correlation between intrathoracic blood volume (ITBV) measured by contrast enhanced ultrasound (CEUS) and magnetic resonance imaging (MRI), as well as the feasibility to use intrathoracic blood volume as a predictor for response to CRT.

Study design: a prospective nonrandomized pilot study Study population: patients with heart failure New York Heart Association (NYHA) class III or IV, a left ventricular ejection fraction equal to or less than 35% and a QRS-duration equal to or more than 0.12 seconds who are referred to our centre for implantation of a CRT-P or CRT-D device.

Intervention: No specific intervention will be performed. Main study parameters: correlation between intrathoracic bloodvolume measured by CEUS and MRI, correlation between LVEF measured by CEUS and by standard 2D ultrasound (biplane methods of discs), change in intrathoracic blood volume as a response to CRT.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: at baseline a clinical examination, laboratory analysis, cardiopulmonary exercise testing, echocardiography and cardiac magnetic resonance imaging will be performed. All of these examinations will be repeated at 3-months follow-up except for the cardiac magnetic resonance imaging. All examinations, except for the MRI, are part of the standard workup in our hospital for patients undergoing implantation of a CRT device. Data needed for the purpose of this study, will be acquired by offline image analysis with dedicated software.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18y
2. LVEF ≤35%
3. QRS-duration ≥0.12 seconds
4. NYHA functional class III or IV despite optimal medical therapy defined as use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor blocker and beta-blockers unless they are not tolerated or contra-indicated
5. sinus rhythm or atrial fibrillation

Exclusion Criteria:

1. episode of acute heart failure ≤3 months
2. change in dosage of beta-blockers, angiotensin-converting enzyme inhibitors or angiotensin-II receptor blockers ≤3 months
3. unstable angina pectoris, acute myocardial infarction, percutaneous intervention or coronary bypass surgery ≤3 months
4. chronic atrial arrhythmias other than atrial fibrillation
5. any mechanical or biological valve prosthesis
6. atrial septal defect
7. right-to-left shunt
8. severe pulmonary hypertension (systolic pulmonary artery pressure >90 mmHg)
9. uncontrolled arterial hypertension
10. known allergy to sulphur hexafluoride
11. end-stage renal or hepatic disease
12. inability to provide written informed consent
13. pregnancy or childbearing potential without use of birth-control measurements
14. general contra-indications to magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to our centre for implantation of a CRT-P or CRT-D device are eligible. In the pilot phase 20 patients will be included. Data will be collected at baseline and 3 months post-implantation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
a. change in ITBV measured by CEUS before and after CRT | two years anticipated
b. correlation of ITBV measured by CEUS and MRI before CRT | two years anticipated

SECONDARY OUTCOMES:
a. correlation between LVEF estimated with CEUS and standard contrast 2D ultrasound | two years anticipated
b. correlation between LVEF estimated with CEUS and MRI | two years anticipated

CONTACTS AND LOCATIONS:
Overall Officials: I.H.F. Herold, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Derived] Herold IH, Saporito S, Mischi M, van Assen HC, Bouwman RA, de Lepper AG, van den Bosch HC, Korsten HH, Houthuizen P. Pulmonary transit time measurement by contrast-enhanced ultrasound in left ventricular dyssynchrony. Echo Res Pract. 2016 Jun;3(2):35-43. doi: 10.1530/ERP-16-0011. Epub 2016 May 16. PMID 27249553